CLINICAL TRIAL: NCT04654533
Title: SEnsitive Care: Understanding and REsponding - Promoting Sensitivity in Center-based Childcare of 0-2 Year Old Children (the SECURE Project)
Brief Title: Promoting Sensitivity in Center-based Childcare
Acronym: SECURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Independent Research Fund Denmark (Industry); TrygFonden, Denmark (Industry); University of Groningen (Other); The Danish Evaluation Institute (Unknown)
Responsible Party: Principal Investigator, Johanne Smith-Nielsen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 514-0151/20-2000
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Caregiver Interactive Skills
Keywords: Quality of care in center-based early childcare

STUDY DESIGN:
Intervention Model Description: Participants are randomized into intervention group or a waitlist
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COSC (Experimental): Eight weekly manualized sessions of Circle of Security Classroom (COSC), delivered in groups, two hours per session, 5-10 childcare providers per group.
  COSC is facilitated by a psychologist who is a registered COSP facilitator and who has completed the an additional COSC online training.
  Interventions: Other: COSC
- Control (No Intervention): Usual care control condition, i.e., standard practice in the participating childcare centers.
  Teams of childcare providers are allocated to either COSC or waitlist in clusters, and baseline and follow-up measures are collected parallel in both groups. Childcare providers allocated to the waitlist will receive COSC after the follow-up data have been collected.

INTERVENTIONS:
Other: COSC — COSC is professional development program for early childcare providers adapted from the Circle of Security-Parenting (COSP) model. It is a manualized intervention that leverages research on attachment relationships combining psycho-education with a mentalization-based approach. The model uses pre-produced video vignettes of secure and problematic caregiver-child interactions to illustrate how caregivers' may struggle in meeting children's' attachment needs.
  Participants are invited to reflect on how they meet and perhaps still not meet the needs of the children in their care with a particular focus on the challenging or 'difficult' children.
  The COSP manual has been translated into Danish (Cooper, Hoffman and Powel, 2020, translated by Pedersen, Kronendorf von Wowern, Lier, & Smith-Nielsen), and the additional COSC material has been translated into Danish for the purpose of this study.
  Arms: COSC

SUMMARY:
The purpose of this study is to test the efficacy of an attachment research-informed intervention adapted to the Danish childcare context in terms of improving process quality in center-based childcare for 0-2 years old children. Specifically, the aim is to improve caregiver interactive skills and mind-mindedness. The intervention is delivered in groups during eight weekly sessions and is based on the manualized Circle of Security Parenting model, but adapted to the childcare context: The Circle of Security Classroom model. Intake is planned to be completed in January 2023 and 110 childcare providers are estimated to be enrolled in the trial.

DETAILED DESCRIPTION:
Background:

It is well-established that children's early attachment relationship experiences with their primary caregivers play an important role in psycho-social development. However, it has been shown that also the child's relationship with other important caregivers, such as early professional caregivers in childcare, is important for socioemotional and academic development. In particular, if a child grows up in an at-risk context the quality of early childcare is pivotal for long-term development.

Children with an insecure attachment to their parents are at heightened risk for developing insecure attachments to professional caregivers. However, caregiver interactive skills are found to be associated with children's attachment security to professional caregivers, irrespective of the child's attachment relationship to the primary caregiver. Therefore, professional caregivers' ability to establish optimal interactions with the children in their care provides an important target of intervention in terms of promoting healthy child development.

In a randomized waitlist control trial, this study aims to

1. investigate the efficacy of COS-C in enhancing caregivers' interactive skills when interacting with groups of children in a natural busy real-life setting, their mind-mindedness (MM), and their work-specific resources to cope with stress.
2. investigate if changes in the caregivers' mind-mindedness is related to changes in their interactive skills.
3. explore if effects of the COS-C are moderated by personal and structural factors, here operationalized as the caregivers' own attachment style and staff stability.
4. evaluate the implementation of the COS-C by examining childcare providers' experience of the intervention's acceptability and feasibility, and we will examine the degree to acceptability and feasibility are related to the intervention's effectiveness. Investigating feasibility and acceptability of the COS-C intervention is essential in terms of evaluating the potential for up-scaling and further implementation of the intervention in Denmark
5. employing a qualitative approach we investigate a) how the caregivers and their managers make sense of changes caused by the intervention and b) how the caregivers experience the intervention in terms of its feasibility and acceptability when implemented in their daily practice.

Methods:

Childcare centers are recruited from a Danish municipality with a high proportion of at-risk families. Teams of 2-5 caregivers working in Danish childcare centers with children aged 0-2 years are allocated to either COS-C (eight weekly two-hour sessions) or a waitlist. A total of 110 caregivers are estimated to be enrolled, and the intervention will be delivered in groups of 6-10 caregivers. To facilitate implementation, the managers of the participating childcare providers are invited to participate in the intervention.

Effects of COS-C are measured using observations of video-recorded caregiver-child interaction (coded for six key interactive skills: Sensitive responsiveness, Respect for autonomy, structuring and limit setting, Verbal communication, Developmental stimulation, and Fostering positive peer interactions) and Mind-Mindedness (representational and interactional Mind-Mindedness) is measured via coding of transcribed interviews and video-recorded caregiver-child interactions. Structural and caregiver attachment style are measured using observation and questionnaires answered by caregivers and managers. Feasibility and acceptability of the intervention are evaluated using questionnaires and via qualitative interviews.

Perspectives:

The project will provide new knowledge on whether a relatively cost-effective intervention can improve the quality of care in Danish childcare centers for young children. Also, findings on how structural factors influence the quality of care will directly inform practice.

ELIGIBILITY:
Inclusion Criteria:

Childcare providers who work in Danish childcare centers ("dagtilbud") for children aged 0 - 60 months in the Municipality of Høje-Taastrup can participate in the study.

Childcare providers with an educational background within childcare as well as childcare providers without education within childcare are included.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Caregiver Interactive Profile (CIP-scales), Sensitive responsiveness scale. | 12-16 weeks
  Coding of sensitive responsiveness is based on video-recorded caregiver-child interactions and sensitivity is rated on a 7-point scale with higher ratings reflecting higher levels of sensitivity

SECONDARY OUTCOMES:
The Mind-Mindedness Interview | 12-16 weeks
  Representational Mind-Mindedness is based on coding of a transcribed brief interview. Each attribute that refers to the child is classified into four categories: 1) Mental attributes, 2) Behavioral attributes, 3) Physical attributes, 4) General attributes, 5) Self-referential comments and 6) Comments regarding institutional practices. The index of representational MM is the total number of mental attributes with higher scores reflecting more Mind-Mindedness.
Interactional Mind-Mindedness | 12-16 weeks
  Coding of interactional Mind-Mindedness is based on observation of video-recorded caregiver-child interaction. Each recording is transcribed verbatim. The transcript is used to identify all mind-related comments that are coded dichotomously as appropriate versus non-attuned by observing the recorded interaction. The two indexes of interactional Mind-Mindedness are: 1) total number of appropriate comments, mind-related, and 2) non-attuned, mind-related comments, with higher scores of appropriate comments reflecting more optimal mind-mindedness and higher scores of non-attuned comments reflecting less optimal mind-mindedness.
Caregiver Interactive Profile (CIP-scales), Respect for autonomy, Structuring and limit setting, Verbal communication, Developmental stimulation, and Fostering positive peer interactions. | 12-16 weeks
  Coding of each interactive skill is based on observation of video-recorded caregiver-child interaction and is rated on a 7-point scale with higher ratings reflecting more optimal interaction.
The Child Care Worker Job Stress Inventory | 12-16 weeks
  The Job resources sub scale is used. 17 questions that are rated on a 5-point likert scale from 1: rarely/never to 5: most of the time.

OTHER OUTCOMES:
The Acceptability of Intervention Measure (AIM) | 12-16 weeks
  3 questions that are rated on a 5-point likert scale ranging from Completely disagree to Completely agree
Feasibility of Intervention Measure (FIM) | Up to 16 weeks
  4 questions that are rated on a 5-point likert scale ranging from Completely disagree to Completely agree.
Client Change Interview. | Up to 16 weeks
  A semi-structured qualitative interview aiming to help clients express (as freely as possible) how they experience a psychotherapeutic intervention has worked. The interview guide has been adjusted to fit the childcare context and the specific intervention for the purpose of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Smith-Nielsen J, Wendelboe KI, Mohr JEW, Vaever MS, Pontoppidan M, Helmerhorst K, Egmose I. Promoting interactive skills and mind-mindedness among early childcare professionals: study protocol for a randomized wait-list controlled trial comparing the Circle of Security approach with care as usual in center-based childcare (the SECURE project). BMC Psychol. 2022 Jun 18;10(1):153. doi: 10.1186/s40359-022-00835-3. PMID 35717243